CLINICAL TRIAL: NCT00586950
Title: Outcome Study on BMIPP SPECT Analysis for Decreasing Cardiac Events in Hemodialysis Patients
Brief Title: 123I-BMIPP SPECT Analysis for Decreasing Cardiac Events in Hemodialysis Patients
Acronym: B-SAFE
Status: Completed | Type: Observational
Sponsor: Translational Research Center for Medical Innovation, Kobe, Hyogo, Japan (Other)
Collaborators: Toho University Ohashi Medical Center (Unknown)
Responsible Party: Kenjiro Kikuchi, MD, PhD , Principal Investigator, Hokkaido Cardiovascular Hospital
Other Study IDs: UHA_CAD05-01
Record Dates: First submitted 2007-12-21; First posted 2008-01-07 (Estimated); Last update posted 2011-09-13 (Estimated); Status verified 2009-02

CONDITIONS: Coronary Disease; Fatty Acids, Unsaturated; Radioisotopes; Hemodialysis; Single Photon Emission Computed Tomography
Keywords: Myocardial Free Fatty Acid metabolism; High risk patients; End-stage renal failure; Cardiovascular events; prognosis
MeSH Terms: conditions — Coronary Disease; Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The aim of this multi-center study is to determine the applicability of BMIPP to diagnosing cardiac disease and to predicting the outcome of patients on hemodialysis.

ELIGIBILITY:
Inclusion Criteria:Adult hemodialysis patients with one or more of the following 10 risk factors for coronary heart disease

* Hypertension
* Diabetes mellitus
* Hyperlipidemia
* Obliterative arteriosclerosis in the lower extremities
* Smoker
* Family history of juvenile coronary artery disease
* History of ischemic stroke
* History of heart failure requiring hospitalization
* Within 3 months after initiation of hemodialysis therapy
* Dialysis hypotension

Exclusion Criteria:Hemodialysis patients who meet any one of the following conditions will be excluded.

* Peritoneal dialysis
* Severe valvular disorder requiring treatment
* Diagnosis of hypertrophic cardiomyopathy(HCM) or dilated cardiomyopathy(DCM) before start of dialysis
* History of revascularization(PCI, CABG) or prior diagnosis of myocardial infarction
* Hypersensitivity to BMIPP or its analogue
* Judged unsuitable for the study for any other reasons by physicians.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Defined Population
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2006-06; Primary Completion 2010-11 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenjiro Kikuchi, MD, PhD, Principal Investigator — Asahikawa Medical College
Locations (1):
- Toho University Ohashi Medical Center, Meguro-ku, Tokyo, Japan